CLINICAL TRIAL: NCT05323734
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled Trial of Adjunctive Ganaxolone (GNX) Treatment in Children and Adults With Tuberous Sclerosis Complex (TSC)-Related Epilepsy (TrustTSC)
Brief Title: Adjunctive GNX Treatment Compared With Placebo in Children and Adults With TSC-related Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1042-TSC-3001
Record Dates: First submitted 2022-03-21; First posted 2022-04-12 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Tuberous Sclerosis Complex-Related Epilepsy; Ganaxolone; Adjunctive
MeSH Terms: conditions — Tuberous Sclerosis | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ganaxolone (GNX) (Experimental): oral suspension, 3 times a day (TID)
  Interventions: Drug: Ganaxolone
- Placebo matching GNX (Placebo Comparator): oral suspension, TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ganaxolone — GNX will be administered
  Arms: Ganaxolone (GNX)
Drug: Placebo — Placebo will be administered
  Arms: Placebo matching GNX

SUMMARY:
This is a Phase 3, global, double-blind, randomized, placebo-controlled study of adjunctive GNX treatment in children and adults with TSC-related epilepsy. The study consists of a 4-week prospective Baseline phase, defined as the first 28 days following screening, followed by a double-blind phase consisting of a 4-week titration period (Day 1 to Day 28) and a 12-week maintenance period (Day 29 to Week 16).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or mutational diagnosis of TSC consistent with:

   1. Molecular confirmation of a pathogenic mutation in TSC1 or TSC2. A pathogenic mutation is defined as a mutation that clearly prevents protein synthesis and/or inactivates the function of the TSC1 or TSC2 proteins (eg, nonsense mutation or frameshift mutations, large genomic deletions) or is a missense mutation whose effect on protein function has been established by functional assessment. The Principal investigator (PI) or designee must review the results of the genetic analysis and confirm that the causal relationship to the epilepsy syndrome is likely. OR
   2. Clinical diagnosis of definite TSC which includes 2 major features or 1 major feature with ≥ 2 minor features.
2. Male or female participants aged 1 through 65 years, inclusive. For Europe (EU), Middle East and North Africa (MENA), and Oceania (OC) Male or Female participants aged 2 through 65 years, inclusive.
3. Participant/parent(s) or LAR(s) willing to give written informed consent/assent, after being properly informed of the nature and risks of the study and prior to engaging in any study related procedures. If the participant is not qualified nor able to provide written informed consent based on age, developmental stage, intellectual capacity, or other factors, parent(s)/LAR(s) must provide consent for study participation, if appropriate.
4. Failure to control seizures despite appropriate trial of 2 or more Anti-seizure medication (ASMs) at therapeutic doses and for adequate duration of treatment per PI judgment.
5. Participants should be on a stable regimen of ASMs (including moderate or strong inducer or inhibitor ASM eg, carbamazepine, phenytoin, etc.) at therapeutic doses for ≥ 28 days prior to the screening visit, and without a foreseeable change in dosing for the duration of the study. (Note: Minor dose adjustment to address tolerability and safety events may be allowed on case-by-case basis and it should be discussed with the study medical monitor.)
6. A history of at least 8 countable seizures per month in the 2 months prior to screening with no more than 1 seizure free week in each month. This includes seizures of any kind.
7. Have at least 8 primary endpoint seizures in the first 28 days following the screening visit.

   The primary endpoint seizure types are defined as the following:
   1. focal motor seizures without impairment of consciousness or awareness
   2. focal seizures with impairment of consciousness or awareness with motor features
   3. focal seizures evolving to bilateral, tonic-clonic seizures
   4. generalized motor seizures including tonic-clonic, bilateral tonic, bilateral clonic, or atonic/drop seizures.

   Seizures that do not count towards the primary endpoint include:
   1. Focal or generalized nonmotor seizures (eg, absence seizures or focal nonmotor seizures with or without impairment of awareness)
   2. Infantile or epileptic spasms
   3. Myoclonic seizures.
8. Participants with surgically implanted vagal nerve stimulator (VNS) will be allowed to enter the study provided that all of the following conditions are met:

   1. The VNS has been in place for ≥ 6 months prior to the screening visit.
   2. The settings must have remained constant for 3 months prior to the screening visit and are expected to remain constant throughout the study.
   3. The battery is expected to last for the duration of the study.
9. Parent(s)/caregiver(s)/LAR(s) or the participant, as appropriate, is (are) willing and able to maintain an accurate and complete daily seizure eDiary for the duration of the study.
10. Willing and able to take IP (suspension) as directed with food (TID).
11. Women of childbearing potential (WOCBP) must be using a medically acceptable method of birth control and have a negative quantitative serum beta-human chorionic growth hormone (β-HCG) test collected at the initial screening and Baseline visits.Childbearing potential is defined as a female who is biologically capable of becoming pregnant. A medically acceptable method of birth control includes intrauterine devices (that have been in place for at least 1 month prior to the screening visit), hormonal contraceptives (eg, combined oral contraceptives, patch, vaginal ring, injectables, and implants), and surgical sterilization (such as oophorectomy or tubal ligation. When used consistently and correctly, "double-barrier" methods of contraception can be used as an effective alternative to highly effective contraception methods. Contraceptive measures such as Plan B™, sold for emergency use after unprotected sex, are not acceptable methods for routine use.
12. Male participants must agree to use highly effective contraceptive methods during the study and for 30 days after the last dose of IP. Highly effective methods of contraception include surgical sterilization (such as a vasectomy) and adequate "double-barrier" methods.

Exclusion Criteria:

1. Previous exposure to GNX.
2. Pregnant or breastfeeding.
3. Participants who have been taking felbamate for less than 1 year prior to screening.
4. Participants taking cannabidiol (CBD) preparations other than Epidiolex.
5. A positive result on plasma drug screen for CBD or tetrahydrocannabinol (THC) at Visit 1 (screening), with the exception of results that are fully explained by Epidiolex, which can be adjusted by the investigator in the event of any Adverse events (AEs).
6. Concurrent use of adrenocorticotropic hormone (ACTH), prednisone or other glucocorticoid is not permitted, nor use of the strong inducers of cytochrome P450 3A4 (CYP3A4), rifampin and St John's Wort. Participants on ACTH, prednisone, or other systemically (non-inhaled or topical) administered steroids should be off the product > 28 days prior to screening. Rifampin and St John's Wort must be discontinued at least 28 days before Visit 2, study drug initiation.

   Note:
   1. Use of concomitant intranasal or pro re nata (PRN) topical steroids for dermatologic reactions and allergic rhinitis are allowed during the study.
   2. This exclusion criterion does not prohibit the use of approved ASMs.
7. Changes in any chronic medications within the 4 weeks prior to the screening visit. All chronic concomitant medications must be relatively stable in dose for at least 4 weeks prior to the screening visit unless otherwise noted. Small dose adjustment to manage tolerability and safety events is permitted and should be discussed with the study medical monitor.
8. Participants who have epilepsy surgery planned during the study or who have undergone surgery for epilepsy within the 6 months prior to screening.
9. An active central nervous system (CNS) infection, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive as evaluated by brain magnetic resonance imaging (MRI). This includes tumor growth which in the opinion of the investigator could affect primary endpoint seizure control.
10. Any disease or condition (medical or surgical; other than TSC) at the screening visit that might compromise the hematologic, cardiovascular (including any cardiac conduction defect), pulmonary, renal, gastrointestinal, or hepatic systems; or other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the IP, or would place the participant at increased risk or interfere with the assessment of safety/efficacy. This may include any illness in the past 4 weeks which in the opinion of the investigator may affect seizure frequency.
11. Hepatic impairment sufficient to affect participant safety, or an aspartate aminotransferase (AST)/ serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SGPT) > 3 × the upper limit of normal (ULN) at screening or Baseline visits and confirmed by a repeat test.
12. Biliary impairment sufficient to affect participant safety, or total bilirubin levels > 1.5 × ULN at screening or Baseline visit and confirmed by a repeat test. In cases of Gilbert's Syndrome, resulting in stable levels of total bilirubin greater than ULN, the medical monitor can determine if a protocol exception can be made
13. Renal impairment sufficient to affect participant safety, or estimated glomerular filtration rate (eGFR) < 30 milliliter per minute (mL/min) (calculated using the Cockcroft-Gault formula or Pediatric GFR calculator or Bedside Schwartz), will be excluded from study entry or will be discontinued if the criterion is met post Baseline. Cases of temporary renal insufficiency should be discussed with the medical monitor to determine the participant's study continuation.
14. Exposed to any other investigational drug or investigational device within 30 days or fewer than 5 half-lives prior to the screening visit. For therapies in which half-life cannot be readily established, the Sponsor's Medical Monitor should be consulted.
15. Unwillingness to avoid excessive alcohol use throughout the study.
16. Have active suicidal plan/intent, active suicidal thoughts or a suicide attempt in the past 6 months.
17. Known sensitivity or allergy to any component in the IP(s), progesterone, or other related steroid compounds.
18. Participants deprived of their liberty by a judicial or administrative decision, or for psychiatric treatment, or participants admitted to a health or social services facility for purposes other than research.
19. Participants receiving traditional Chinese medicine therapies within the prior 28 days of the screening.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (23):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - UCLA Mattel Children's Hospital, TSC Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Diego, San Diego, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital - Delaware Valley, Wilmington, Delaware
  - University of Florida Gainesville, Gainesville, Florida
  - Nemours Children's Health, Jacksonville, Florida
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Children's Mercy Hosptial, Kansas City, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health/Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Child Neurology Consultants of Austin (CNCA), Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - McGovern Medical School at the University of Texas Health Science Center, Houston, Texas
  - University of Utah Health Care-Pediatric Neurology, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Austin Health, Heidelberg
  - Alfred Health, Melbourne
  - Royal Melbourne Hospital, Parkville
- Canada (5):
  - Hôtel Dieu de Montréal - CHUM, Montreal
  - CHU Sainte-Justine, Montreal
  - The Hospital for Sick Children, Toronto
  - Toronto Western Hospital, Toronto
  - BC Children's Hospital, Vancouver
- China (7):
  - First Hospital of Jilin University, Changchun, Jilin
  - Jiangxi Provincial Children's Hospital, Jiangxi, Nanchang City
  - Beijing Children Hospital, Capital Medical University, Beijing, Xicheng District
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Yunyan District
  - Peking University First Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Chengdu's Women and Children's Central Hospital, Chengdu
- France (3):
  - University Hospital of Lyon, Bron
  - University Hospital of Rennes, Rennes
  - University of Strasbourg, Strasbourg
- Germany (6):
  - Epilepsie-Zentrum Bethel - Krankenhaus Mara, Bielefeld
  - University Hospital Bonn, Bonn
  - ZNN - Epilepsiezentrum Frankfurt am Main, Frankfurt
  - Universitäts Krankenhaus Freiburg, Freiburg im Breisgau
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - Epilepsiezentrum Kleinwachau gGmbH, Radeberg
- Israel (2):
  - Schneider Children´s Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Department of Neurology and Sense Organs, AOU Policlinico di Bari, Bari
  - Pediatric Neurology and Muscular Diseases Unit - University of Genoa, Genova
  - Policlinico Umberto I, Rome
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Ruber International, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (4):
  - Bristol Royal Hospital for Children, Bristol
  - NHS acute tertiary referral centre, John Radcliffe Hospital, Oxford
  - Salford Royal Hospital, Salford
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, global, double-blind, randomized, placebo-controlled study of adjunctive Ganaxolone treatment in children and adults with TSC-related epilepsy.
Pre-assignment Details: A total of 129 participants were enrolled in the study.
Groups:
- Ganaxolone: Participants were randomized to receive an oral suspension of Ganaxolone based on their body weight. Ganaxolone 63 milligrams/kilograms/day (mg/kg/day) was administered orally three times a day (TID) to participants weighing 28 kg or less. Ganaxolone 1800 mg/day TID was administered orally to participants weighing more than 28 kg.
- Placebo: Participants were administered with matching placebo as oral suspension TID based on the body weight.
Period: Overall Study
Arm/Group | Ganaxolone | Placebo
Started | 64 | 65
Completed | 55 | 60
Not Completed | 9 | 5
Not completed — Adverse Event | 5 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Participant Withdrawn Due | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set comprised of all randomized participants who receive at least 1 dose of the investigational product (IP).
Groups:
- Matching Placebo: Participants were administered with matching placebo as oral suspension TID based on the body weight.
- Total: Total of all reporting groups
Arm/Group | Ganaxolone | Matching Placebo | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.7 (11.0) | 16.1 (11.2) | 15.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 28 | 36 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 52 | 55 | 107
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 11 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 41 | 48 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 28-day Seizure Frequency for Primary Seizure Type During Double Blind Period
Description: Primary seizures include atonic/drop, bilateral clonic, bilateral tonic, focal motor with altered awareness, focal motor with intact awareness, focal to bilateral tonic-clonic seizures, focal with hypotonia impaired awareness, and generalized tonic-clonic. Seizure frequency was calculated as the total number of seizures divided by the number of days with seizure data in the period, multiplied by 28. Percent change from Baseline in 28-day seizure frequency was calculated as follows for each participant: post-baseline 28-day seizure frequency minus baseline 28-day seizure frequency whole divided by baseline 28-day seizure frequency and multiplied by 100.
Time Frame: Baseline (Day 1), Day 28
Population: Intent-to-treat (ITT) Set comprises of randomized participants who dosed and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Ganaxolone: Participants were randomized to receive oral suspension of Ganaxolone 63 milligrams/kilograms/day (mg/kg/day) for those weighing 28 kg or less and 1800 mg/day for those weighing more than 28 kg three times a day.
- Matching Placebo: Participants were administered with matching placebo as oral suspension 3 times a day.
Arm/Group | Ganaxolone | Matching Placebo
Number analyzed (Participants) | 64 | 65
Percent change | -7.50 (60.430) | 13.57 (77.374)
Statistical Analysis 1: Comparison: Ganaxolone vs Matching Placebo; Test type: Other; p = 0.0904, Wilcoxon Rank-Sum; Wilcoxon Rank-Sum statistic is applied using a 2-sided significance level of 0.05; Median Difference (Final Values) = -14.53, 95% CI 2-sided [-32.04 to 2.48] — The Hodges-Lehmann approach is applied for estimating 95% confidence interval

2. Secondary Outcome: Number of Participants Who Were Considered as Treatment Responders During Double Blind Period
Description: Treatment responders are defined as those participants with ≥ 50% reduction from Baseline in primary seizure type frequency during the given period.
Time Frame: Up to 16 weeks
Population: ITT Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Matching Placebo
Number analyzed (Participants) | 64 | 65
Participants | 12 | 8
Statistical Analysis 1: Comparison: Ganaxolone vs Matching Placebo; Test type: Other; p = 0.3407, Fisher Exact; Difference in percentage = 6.4, 95% CI 2-sided [-6.4 to 20.1]

3. Secondary Outcome: Number of Responders to Clinical Global Impression of Improvement (CGI-I) Scale as Assessed by Parent/Caregiver
Description: The CGI-I is a 7-point Likert scale that the parent(s)/caregiver(s)/ legally authorized representative (LAR) and clinician uses to rate the change in overall seizure control, behavior, safety, and tolerability after initiation of the IP relative to baseline (prior to treatment with the IP). The participant was rated as follows: 1 - very much improved, 2 - much improved, 3 - minimally improved, 4 - no change, 5 - minimally worse, 6 - much worse, and 7 - very much worse. Higher scores indicated worse condition. Number of responders to each score on the scale has been presented.
Time Frame: Baseline (Day 1) through 16 weeks
Population: ITT Set. Only those participants who responded to CGI-I scale has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Matching Placebo
Number analyzed (Participants) | 58 | 58
Participants
  Very Much Improved | 5 | 8
  Much Improved | 16 | 15
  Minimally Improved | 14 | 12
  No Change | 19 | 19
  Minimally Worse | 2 | 4
  Much Worse | 2 | 0
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Ganaxolone vs Matching Placebo; Test type: Other; p = 0.7069, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.46 to 1.70] — The estimated odds ratio of the ganaxolone group compared to the placebo group based on proportional odds logistic regression with treatment as a factor

4. Secondary Outcome: Number of Responders to Clinical Global Impression of Improvement (CGI-I) Scale as Assessed by Clinician
Description: The CGI-I is a 7-point Likert scale that the parent(s)/caregiver(s)/ LAR and clinician uses to rate the change in overall seizure control, behavior, safety, and tolerability after initiation of the IP relative to baseline (prior to treatment with the IP). The participant was rated as follows: 1 - very much improved, 2 - much improved, 3 - minimally improved, 4 - no change, 5 - minimally worse, 6 - much worse, and 7 - very much worse. Number of responders to each score on the scale has been presented.
Time Frame: Baseline (Day 1) through 16 weeks
Population: ITT Set. Only those participants who responded to CGI-I scale has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Matching Placebo
Number analyzed (Participants) | 51 | 53
Participants
  Very Much Improved | 0 | 3
  Much Improved | 14 | 13
  Minimally Improved | 12 | 11
  No Change | 22 | 25
  Minimally Worse | 2 | 1
  Much Worse | 1 | 0
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Ganaxolone vs Matching Placebo; Test type: Other; p = 0.6434, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.42 to 1.72] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 16 Weeks
Description: Serious treatment emergent adverse events and treatment emergent adverse events were collected in Safety Analysis Set which comprises of all randomized participants who received at least 1 dose of the IP.
Arm/Group | Ganaxolone | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/65
Serious Adverse Events (participants affected / at risk) | 5/64 | 6/65
Other Adverse Events (participants affected / at risk) | 58/64 | 49/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=64) | Matching Placebo (N=65)
Erysipelas (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia Aspiration (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=64) | Matching Placebo (N=65)
Somnolence (Nervous system disorders) | 18 | 11
Seizure (Nervous system disorders) | 9 | 8
Headache (Nervous system disorders) | 6 | 2
Balance Disorder (Nervous system disorders) | 3 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 3 | 0
Sedation (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 5 | 4
Influenza (Infections and infestations) | 4 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 6
Conjunctivitis (Infections and infestations) | 2 | 1
Covid-19 (Infections and infestations) | 2 | 3
Respiratory Tract Infection (Infections and infestations) | 2 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Mouth Ulceration (Gastrointestinal disorders) | 3 | 1
Dental Caries (Gastrointestinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 10 | 11
Fatigue (General disorders) | 9 | 6
Asthenia (General disorders) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3
Skin Abrasion (Injury, poisoning and procedural complications) | 2 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 4
Increased Appetite (Metabolism and nutrition disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Affect Lability (Psychiatric disorders) | 2 | 0
Irritability (Psychiatric disorders) | 2 | 4
Sleep Disorder (Psychiatric disorders) | 2 | 3
Aggression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 2
Weight Increased (Investigations) | 3 | 0
Weight Decreased (Investigations) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Menstruation Irregular (Reproductive system and breast disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT05323734/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT05323734/SAP_001.pdf